CLINICAL TRIAL: NCT06032455
Title: The Effectiveness of Multisystemic Therapy for Adolescents With Severe Behavioural Problems From Families With Intellectual Disabilities: A Mixed-Method Study
Brief Title: Effectiveness of Multisystemic Therapy for Adolescents From Families With Intellectual Disabilities
Status: Recruiting | Type: Observational
Sponsor: De Viersprong (Other)
Collaborators: Stichting tot Steun (Unknown); Koraal (Other); Prisma (Unknown); MST-Netherlands/Belgium (Unknown); Radboud University Medical Center (Other); Pactum (Unknown)
Responsible Party: Sponsor
Other Study IDs: 303
Record Dates: First submitted 2023-07-25; First posted 2023-09-13 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-06

CONDITIONS: Behavioural Problems
Keywords: multisystemic therapy; intellectual disability; adolescent behavioural problems; family functioning
MeSH Terms: conditions — Mental Disorders; Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Families receiving standard MST: Families in which the adolescent and/or parent(s) has/have an ID receiving standard MST treatment
  Interventions: Behavioral: Multisystemic therapy
- Families receiving MST-ID: Families in which the adolescent and/or parent(s) has/have an ID receiving MST-ID treatment
  Interventions: Behavioral: Multisystemic therapy - intellectual disabilities

INTERVENTIONS:
Behavioral: Multisystemic therapy — Multisystemic Therapy (MST) is an intensive, evidence-based treatment aimed at preventing out-of-home placement of adolescents with severe behavioural problems. The intervention is home-based and focuses not only on the adolescent, but also on the various systems surrounding the adolescent, such as the family, neighbourhood, school, and friends. MST helps parents increase their parenting competencies such as parental monitoring and find (more) social support in their environment. MST also helps adolescents improve their relationship with their parents, school participation, and social activities, and promotes contact with pro-social peers. These goals are achieved by working together with key figures in the family's environment. MST treatment duration is three to five months. In MST, a family can contact a therapist 24/7.
  Other Names: MST
  Groups: Families receiving standard MST
Behavioral: Multisystemic therapy - intellectual disabilities — Multisystemic therapy - intellectual disabilities (MST-ID) is a specialisation of standard MST (see above), tailored to the needs and skill deficits of families in which the adolescent and/or parent(s) has/have a known or suspected ID. In MST-ID, among others, simplified language and visual support are used, and extra attention is paid to the generalisation of what has been learned in the treatment sessions.
  Other Names: MST-ID
  Groups: Families receiving MST-ID

SUMMARY:
The goal of this observational study is to determine the effectiveness of a specialisation of multisystemic therapy (MST) for adolescents with severe behavioural problems from families with an intellectual disability (ID; MST-ID).

To achieve this goal, a mixed method study design is used. To this end, a quantitative and a qualitatively primary research question are formulated:

* Is MST-ID superior, when compared to standard MST, in reducing rule-breaking behaviour of adolescents (quantitative)?
* What are the experiences of adolescents and/or parents receiving MST-ID treatment (qualitative)?

Participants will be asked to complete two screeners (questionnaires delivered as a verbal interview) with a total duration of approximately 30 minutes. Other data will be collected through Routine Outcome Monitoring questionnaires that are part of standard MST procedures. To this end, five 'time points' have been identified: T0 (start of MST[-ID] treatment), T1 (end of MST[-ID] treatment), T2 (follow-up 6 month after MST[-ID] treatment), T3 (follow-up 12 month after MST[-ID] treatment), and T4 (follow-up 18 month after MST[-ID] treatment). The qualitative method used to gain insight into families' experiences is determined in consultation with the families.

To assess the effectiveness of MST-ID, its treatment outcomes will be compared to standard MST treatment outcomes of families with ID.

DETAILED DESCRIPTION:
Background of the study:

Over the years, a large body of research has shown that adolescents with intellectual disability are 3-4 times more likely to develop severe behaviour problems than adolescents without intellectual disability. Families in which adolescents and/or one or both parent(s) have an intellectual disability (from now on, families with ID) often deal with complex problems, putting the adolescent at an increased risk of out-of-home placement. Multisystemic therapy (MST) is an intensive home-based treatment, effective in reducing severe behaviour problems and preventing the out-of-home placement of adolescents. A specialisation of MST has been developed for families with ID: MST-ID. In MST-ID, among other alterations, simplified language and visual support is used, sessions are more structured and more time is scheduled for practicing exercises, and extra attention is paid to the generalisation of what has been learned in the sessions (with the aim of attaining long-term outcomes). Pilot studies show that when compared to standard MST, MST-ID shows similar or better treatment outcomes in families with adolescents with ID. Meanwhile, MST-ID has been disseminated more widely and the target population extended by including families in which only the parent(s) have an ID.

Objective of the study:

The aim of this study is to investigate the effectiveness of MST-ID for adolescents with severe behavioural problems from families with an intellectual disability (ID), compared to standard MST. It is hypothesised that MST-ID is more effective - in terms of fewer behavioural problems, more adolescents living at home, being in school/work, no new police contacts, less parenting stress - than standard MST. Treatment outcomes are considered both quantitatively and qualitatively.

Study design:

Quantitatively, the Propensity Score (PS) method is used to balance treatment groups and, combined with Multilevel Modelling (MLM), to estimate treatment effect over time. Qualitatively, the experiences of approximately 10 adolescents and/or parents are centralised. The qualitative research methods will be decided upon in a participatory manner with respondents (examples of potential research methods are interviews, focus group discussions, or photo elicitation).

Study population:

Adolescents (10-19y) with severe behavioural problems or delinquent behaviours, and their parent(s) receiving MST(-ID) treatment. All research participants must be from families where either the adolescent and/or parent(s) has/have ID.

Intervention:

Following standard referral procedures, families were either referred to standard MST or MST-ID treatment (i.e., non-randomly). Both standard MST and MST-ID are intensive, home-based treatments with 3-5 home visits per week, targeting the severe behavioural problems of adolescents across multiple life domains. MST-ID is tailored to the needs and skill deficits of adolescents and/or parents with ID. Concretely, more attention is paid to how therapists create engagement, implement interventions, and realise support from informal supports, in a tailored, developmentally appropriate, and simplified manner (meaning in a more structured way and using accessible language, among others), when compared to standard MST.

Research questions:

Building on the objectives, the following research questions were formulated:

Primary research questions:

1. Is MST-ID superior, when compared to standard MST, in reducing rule-breaking behaviour of adolescents, according to parents?
2. Is MST-ID superior, when compared to standard MST, in reducing rule-breaking behaviour of adolescents, according to adolescents?

   Secondary research questions:
3. Is MST-ID superior, when compared to standard MST, in reducing externalising and internalising behavioural problems of adolescents, according to parents?
4. Is MST-ID superior, when compared to standard MST, in reducing externalising and internalising behavioural problems of adolescents, according to adolescents?
5. Is MST-ID superior, when compared to standard MST, in reducing parenting stress?
6. Is MST-ID superior, when compared to standard MST, in preventing short and long term out-of-home placement, delinquency, truancy or joblessness, and addictions of adolescents?
7. Is MST-ID superior, when compared to standard MST, in realising improvements on family's social networks?
8. Is MST-ID superior, when compared to standard MST, in improving the instrumental outcome parenting skills?
9. Is MST-ID superior, when compared to standard MST, in improving the instrumental outcome family relations?
10. Is MST-ID superior, when compared to standard MST, in improving the instrumental outcome social support?
11. Is MST-ID superior, when compared to standard MST, in improving the instrumental outcome adolescent success in an educational or vocational setting?
12. Is MST-ID superior, when compared to standard MST, in improving the instrumental outcome adolescent involvement with pro-social peers?
13. Is MST-ID superior, when compared to standard MST, in improving the instrumental outcome change in adolescent problem behaviour?
14. What are the experiences of adolescents and/or parents receiving MST-ID treatment?
15. Do effects across subgroups of adolescents and/or parents with ID differ?

MST-ID is expected to be superior in achieving the aforementioned outcomes (#1-13) when compared to standard MST. Research questions #14-15 will be assessed exploratively, therefore no hypotheses have been formulated.

ELIGIBILITY:
Referral Criteria:

* Known or suspected ID of the referred adolescent and/or their parent(s);
* Educational level of the referred adolescent and/or highest attained diploma of their parent(s) is indicative of potential ID.

Inclusion Criteria Study Sample:

* Adolescent must be 10 to 19 years old at the start of treatment;
* Adolescent presents with severe behavioural problems in at least two life areas;
* Adolescent lives with a family or there is a family the adolescent can live with, in which parent(s) have parental custody for a longer period of time;
* Parent(s) consent(s) and is/are willing to engage in treatment to prevent an out-of-home placement of the adolescent;
* Adolescent and/or parent(s) have a known or suspected intellectual disability (operationalised as an intelligence quotient [IQ] score of between 50-85 and additional deficits in adaptive functioning)
* Adolescent and/or parent(s) have sufficient knowledge of the Dutch language (as assessed by a clinician and/or researcher) in order to understand and answer the various (self-report) questionnaires.

Exclusion Criteria Study Participation:

* Adolescent lives independently;
* Adolescent presents with severe problematic sexual behaviours, without presenting with other severe behavioural problems;
* Adolescent presents suicidal, psychotic, or homicidal requiring specialised treatment (such as a crisis placement in a residential facility);
* Adolescent has a severe Autism Spectrum Disorder (level 2-3 according to the Diagnostic and Statistical Manual of Mental Disorders [DSM-V] criteria) or a severe ID (IQ score <50);
* Adolescent has internalising psychiatric problems which are the primary reason for referral, or has serious psychiatric problems (similar to #3 as well as for example eating disorder.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The target population consists of adolescents and their parent(s) with a known or suspected ID referred to MST-ID at one of three Dutch mental health care organisations (de Viersprong, Koraal, and Prisma) or to standard MST at one of two Dutch mental health care organisations (de Viersprong and Pactum).
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rule-breaking behaviour of adolescents - parents | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  Rule-breaking behaviour of adolescents according to parents will be assessed using the Child Behavior Check List (CBCL). The CBCL consists of 118 questions rated on a 3-point scale from 0 (absent) to 2 (occurs often). Higher scores indicate that adolescents experience more problems.
Rule-breaking behaviour of adolescents - adolescents | Start (T0) and end (T1) of MST(-ID) treatment, an average of 4 months in between
  Rule-breaking behaviour of adolescents according to parents will be assessed using the Youth Self Report (YSR). The YSR consists of 112 questions rated on a 3-point scale from 0 (absent) to 2 (occurs often). Higher scores indicate that adolescents experience more problems.

SECONDARY OUTCOMES:
Externalising and internalising behavioural problems of adolescents - parents | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  Externalising and internalising behavioural problems of adolescents will be assessed using the Child Behavior Check List (CBCL). The CBCL consists of 118 questions rated on a 3-point scale from 0 (absent) to 2 (occurs often). Higher scores indicate that adolescents experience more problems.
Externalising and internalising behavioural problems of adolescents - adolescents | Start (T0) and end (T1) of MST(-ID) treatment, an average of 4 months in between
  Externalising and internalising behavioural problems of adolescents according to adolescents will be assessed using the Youth Self Report (YSR). The YSR consists of 112 questions rated on a 3-point scale from 0 (absent) to 2 (occurs often). Higher scores indicate that adolescents experience more problems.
Parenting stress | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  Parenting stress will be assessed using the Parenting Stress Questionnaire (PSQ). The PSQ consists of 34 questions rated on a 4-point scale from 1 (not true) to 4 (very true). Higher scores indicate more parenting stress.
Out-of-home placement | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  Out-of-home placement of adolescents will be assessed using the Social Demographic Information 3.0 questionnaire (SDI 3.0).
Delinquency | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  Delinquency of adolescents is operationalized as police contact and will be assessed using the SDI 3.0.
School going or work | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  The adolescent's school going or work is operationalised as "school going that meets the expectations of the school or public education law officer or work that meets the expectations of caregivers and the referring agent" and will be assessed using the SDI 3.0.
Addictions | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  Addictions of adolescents are operationalised as "adolescent drug misuse/abuse, screen or game dependency that has resulted in addiction, and/or other addictions" and will be assessed using the SDI 3.0.
Social network | Start of MST(-ID) treatment (T0) until 18-month follow up (T4)
  Social network is operationalised as "forms of social network available to a family and number of supports (read: individuals) that are available to the family" and will be assessed using the SDI 3.0.
IO Percentage of families with improved parenting skills | End of MST(-ID) treatment, an average of 4 months after start of treatment
  MST's so called "instrumental outcomes" (IOs) identify skills which are instrumental to achieving positive treatment outcomes and are reported by therapists. The first IO assesses whether or not families show improved parenting skills, answered 'yes' or 'no'.
IO Percentage of families with improved family relations | End of MST(-ID) treatment, an average of 4 months after start of treatment
  MST's so called "instrumental outcomes" (IOs) identify skills which are instrumental to achieving positive treatment outcomes and are reported by therapists. The second IO assesses whether or not families show improved family relations, answered 'yes' or 'no'.
IO Percentage of families with improved social support | End of MST(-ID) treatment, an average of 4 months after start of treatment
  MST's so called "instrumental outcomes" (IOs) identify skills which are instrumental to achieving positive treatment outcomes and are reported by therapists. The third IO assesses whether or not families show improved social support, answered 'yes' or 'no'.
IO Percentage of families with adolescent success in an educational or vocational setting | End of MST(-ID) treatment, an average of 4 months after start of treatment
  MST's so called "instrumental outcomes" (IOs) identify skills which are instrumental to achieving positive treatment outcomes and are reported by therapists. The fourth IO assesses whether or not the adolescent obtained success in an educational or vocational setting, answered 'yes' or 'no'.
IO Percentage of families with adolescent involvement with pro-social peers | End of MST(-ID) treatment, an average of 4 months after start of treatment
  MST's so called "instrumental outcomes" (IOs) identify skills which are instrumental to achieving positive treatment outcomes and are reported by therapists. The fifth IO assesses whether or not the adolescent is involved with pro-social peers, answered 'yes' or 'no'.
IO Percentage of families with change in adolescent problem behaviour | End of MST(-ID) treatment, an average of 4 months after start of treatment
  MST's so called "instrumental outcomes" (IOs) identify skills which are instrumental to achieving positive treatment outcomes and are reported by therapists. The sixth IO assesses whether or not the adolescent obtained changes in problem behaviour that were sustained for 3-4 weeks, answered 'yes' or 'no'.

OTHER OUTCOMES:
Family and treatment characteristics | Start of MST(-ID) treatment (T0)
  Characteristics of families that are gathered are previous treatment, referral stream and the following:
  Adolescent: age, gender identity, cultural background, prior residential placement, living situation, level of education Primary caregiver: level of education, employment status, partner, experienced financial stress, experienced living situation stress
Intellectual functioning | Start of MST(-ID) treatment (T0)
  Intellectual functioning will be assessed using the Dutch Screener for Intelligence and Learning Disabilities (SCIL). The SCIL consists of 14 questions that result in a total SCIL score that can range from 0 to 28. A total SCIL score of 19 and below indicates the presence of intellectual disabilities.
Adaptive functioning | Start of MST(-ID) treatment (T0)
  Adaptive functioning will be assessed using the Dutch Screener for Adaptive Functioning and Learning Disabilities (SCAF). The SCAF consists of 12 questions that result in a total SCAF score that can range from 0 to 13. A higher score indicates a higher level of adaptive functioning.
Treatment fidelity | Monthly throughout MST(-ID) treatment, an average of 4 months
  Treatment fidelity is measured and checked through administration of a validated questionnaire to the primary caregiver of each family (TAM-R).
Subgroups of ID families | Start of MST(-ID) treatment (T0)
  Families included in this study are divided across three subsamples: families in which only the adolescent, only the parent(s), and both the adolescent and parent(s) have ID. This This variable will be calculated based on participants' SCIL scores.
Experiences of families receiving MST-ID | Through study completion, an average of 1 year
  Experiences of families receiving MST-ID will be assessed using participatory and qualitative research methods. The aim is to recruit 10 adolescents or parents and to ask them to help identify which elements of MST-ID are most important to them, and which elements were found least and most helpful. This can lead to a better understanding of what works well and less well in MST-ID treatments. Potential qualitative research methods are focus group discussions, peer-interviewing, and photo-elicitation/photo voice.

CONTACTS AND LOCATIONS:
Overall Officials: Dineke Feenstra, PhD, Principal Investigator — De Viersprong
Locations (4):
- Netherlands (4):
  - De Viersprong, Halsteren
  - Koraal, Sittard
  - Stichting Prisma, Waalwijk
  - Pactum, Zetten

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emerson E, Einfeld S, Stancliffe RJ. Predictors of the persistence of conduct difficulties in children with cognitive delay. J Child Psychol Psychiatry. 2011 Nov;52(11):1184-94. doi: 10.1111/j.1469-7610.2011.02413.x. Epub 2011 Apr 19. PMID 21501168
- [Background] Blankestein A, van der Rijken R, Eeren HV, Lange A, Scholte R, Moonen X, De Vuyst K, Leunissen J, Didden R. Evaluating the effects of multisystemic therapy for adolescents with intellectual disabilities and antisocial or delinquent behaviour and their parents. J Appl Res Intellect Disabil. 2019 May;32(3):575-590. doi: 10.1111/jar.12551. Epub 2019 Jan 8. PMID 30620111
- [Background] Blankestein A, Lange A, van der Rijken R, Scholte R, Moonen X, Didden R. Brief report: Follow-up outcomes of multisystemic therapy for adolescents with an intellectual disability and the relation with parental intellectual disability. J Appl Res Intellect Disabil. 2020 May;33(3):618-624. doi: 10.1111/jar.12691. Epub 2019 Dec 28. PMID 31883357
- [Background] De Ruiter KP, Dekker MC, Douma JCH, Verhulst FC, Koot HM. Development of parent- and teacher-reported emotional and behavioural problems in young people with intellectual disabilities: Does level of intellectual disability matter? J Appl Res Intellect Disabil. 2008; 21(1): 70-80.
- [Background] Wallander JL, Dekker MC, Koot HM. Psychopathology in children and adolescents with intellectual disability: Measurement, prevalence, course, and risk. International Review of Research in Mental Retardation. 2003; 26: 93-134.
- [Background] Blankestein A, Van der Rijken R, De Vuyst K, De Bruijn J, Moonen X, Leunissen J, Didden R. Multisysteemtherapie voor jongeren met een licht verstandelijke beperking en hun ouders: Een onderzoek naar de effectiviteit van een ambulante systeemgerichte interventie. Directieve Therapie. 2016; 36(3): 204-219. Dutch.
- [Background] Dekker MC. Short Review: Psychopathology in young people with mild ID or borderline intellectual functioning: Research findings from representative (clinical) samples & future needs. Academische Werkplaats Kajak. 2019.
- [Background] Henggeler SW, Schoenwald SK, Borduin CM, Rowland MD, Cunningham PB. Multisystemic therapy for antisocial behavior in children and adolescents. 2nd ed. New York: The Guilford Press; 2009.
- [Background] Kaal HL, Overvest N, Boertjes MJ. Beperkt in de keten: Mensen met een licht verstandelijke beperking in de strafrechtsketen [People with mild intellectual disability in the justice system]. 2nd ed. Amsterdam: Boom Lemma; 2014.